CLINICAL TRIAL: NCT02103868
Title: Interventional Study to Determine the Effectiveness of Medium Intensity Verses Low Intensity Tobacco Use Prevention and Cessation Intervention in the Unorganized Sector of Zari Workers in Mumbai
Brief Title: Medium Vs Low Intensity Intervention in Tobacco Cessation and Control in Zari Workers
Acronym: ZARI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Sharmila Pimple, Professor in Preventive Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: TMHPOZariW2013
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Tobacco Cessation
Keywords: Tobacco cessation; Zari worker; Behavior therapy; Qualitative Research; Mumbai
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): No active intervention will be given for tobacco cessation.
- Medium Intervention (Experimental): Tobacco Cessation Counseling : Medium intervention in the form of 3 contact sessions will be given for tobacco cessation.
  Interventions: Behavioral: Tobacco Cessation Counseling
- Low intensity intervention (Experimental): Tobacco Cessation Counseling: Only a single contact session will be done for tobacco cessation.
  Interventions: Behavioral: Tobacco Cessation Counseling

INTERVENTIONS:
Behavioral: Tobacco Cessation Counseling — Doing group and personal counseling for tobacco cessation
  Other Names: TCC
  Arms: Low intensity intervention; Medium Intervention

SUMMARY:
Zari workers in Mumbai city will be assessed for tobacco consumption habit. They will be divided into 3 arms as - 1) First arm will get Medium intensity tobacco cessation intervention 2) Second arm will get low intensity tobacco cessation intervention 3) Control arm. At the end of 12 months of intervention quit rates will be compared.

DETAILED DESCRIPTION:
Aims and Objectives

Broad objective:

The proposed study is planned to understand prevalence and practices related to tobacco use among workers of the informal sector of Zari Industry and to assess the feasibility and acceptability of effective strategies of a programmatic approach towards tobacco use prevention and cessation intervention model in this by assessment of pre and post-intervention knowledge, attitude and perception of tobacco use, followed by offering education and cessation and finally assessing the impact and outcomes by changes in the attitudes towards tobacco use and quit rates among tobacco users.

Specific objectives:

Primary Objectives:

1. To assess knowledge and understand the practices related to tobacco use among the Zari workers' population using qualitative research.
2. To implement a multicomponent community-based intervention model through trained health workers in an unorganized workplace setting.
3. To assess any change in the Knowledge Attitude and Practices related to tobacco use at post intervention.
4. Determine tobacco cessation rates at the end of intervention.

Secondary Objectives:

1. To provide oral screening service to the target groups at the end of the interventions.
2. Develop a LOCAL -language tobacco use prevention and cessation training module to train counsellors in tobacco cessation interventions.

Study Methodology

Design:

A prospective, community-based randomized controlled design

Settings: Community based Zari work units of three urban slum pockets in Mumbai

Sampling:

Three distinct urban slum communities in Mumbai where Zari units operate will be identified. Each of the slum community will serve as three arms of the trial, with one geographic cluster / community serving as the intervention community for moderate intensity intervention, second cluster /community for low intensity intervention and the third cluster/community serving as the control arm with no intervention. These communities will be recruited on the basis of comparable socio-demographic characteristics.

Tools of Data Collection:

Questionnaire:

A pre designed structured baseline questionnaire will be prepared to understand the determinants that trigger the onset of tobacco use, dynamics of regular use of tobacco and factors that motivate the user to quit tobacco. Written informed consent will be taken from all the participants.

The questionnaire at baseline will be administered in local language before the implementation of the intervention and will be repeated after 1 year with the same sample at end to assess the efficacy of the intervention. The questionnaire will be administered by a trained interviewer as per the convenience of the respondents.

Intervention Arm:

Intervention A community-based multi-component intervention model developed, will be implemented and evaluated in the intervention community. The intervention model will address numerous socio-environmental and intra-personal factors that trigger the onset of tobacco use and other determinants that influence tobacco cessation.

The intervention consists of :

1. Awareness & Education on Tobacco use prevention:

   Interactive activities, pre-tested posters, in addition, pictorial handouts, booklets and pamphlets will be distributed for knowledge enhancement by trained social workers. The first interaction with the workers will involve an elaborate common education programme on harms of tobacco use, tobacco use prevention and benefits of tobacco cessation, by an audio visual presentation and distribution of pamphlets for knowledge enhancement by trained social workers. All participants will be assessed for their tobacco use status prior to the intervention. The participants with history of current tobacco use in any form will then be enrolled for further interventions for tobacco cessation. A structured questionnaire detailing information on sociodemographic variables with medical and other risk factors with complete assessment of their tobacco habit will be entered by medical social workers. All participants will be assessed for their tobacco use status at all interventions.
2. Focus Group discussion:

   This tobacco cessation intervention session with the tobacco users after three months of the first contact program will involve thirty minutes of focus group discussion with group behavioral therapy in groups of 5-10 individuals for reinforcement of tobacco use prevention and cessation advice. Group discussion is intended to improve understanding by exploring, sharing and reflecting psychosocial, familial, environmental issues which attribute to the problem. Members of the group are encouraged to exchange information and ideas about the perceived barriers towards tobacco cessation. Techniques like reflecting, exploring and re-evaluation will be used to identify their problem to improve insight and reinforce attitudinal change.
3. Individual tobacco cessation counseling sessions:

Iindividual counseling is commonly used to help people who are trying to quit tobacco. The counseling adopting a interactive problem-solving approach will be done by trained Medical Social Workers providing face-to-face sessions for 10-15 minutes per participant,

Types of Intervention

1. Medium Intensity Intervention

   The Medium intensity arm will implement the multi-component program with three contact programs.

   I. First Contact program: Group health education session II. Second Contact program: Focus Group Discussion III. Third Contact program: Brief Individual Counseling session
2. Low Intensity Intervention

Single contact session with Group health education session will be provided to the participants

Final Outcome Final outcome measure, the quit rates as self reported tobacco abstinence will be assessed at the end of one year.

Oral cancer screening:

All the Zari workers will also be invited for oral cancer screening at the end of intervention program.

Oral cancer screening to detect clinically recognizable precancerous lesions (leukoplakia, erythroplakia and oral submucous fibrosis) and asymptomatic early invasive lesions will be done by trained Primary Health Workers. Visual examination of the oral cavity with good light source like halogen flashlight, is a simple approach to detect asymptomatic oral cancers and precancerous lesions. The performance characteristics of this test are satisfactory in terms of sensitivity, specificity, and predictive value therefore, it is a suitable screening test for oral cancer. One large study from Kerala has shown that screening by visual inspection of the mouth by trained health workers may potentially reduce mortality in high risk groups.

The clinical findings will be recorded as 1. Normal; 2. Benign or non cancerous lesions such as fissures in the tongue, aphthous ulcer, black patch, tobacco-related blanching, fibroma, hypertrophied papillae, etc.; and 3. Pre cancer lesions if found to have a white patch, ulcerated white patch, verrucous lesion, submucous fibrosis, red patch, suspicious ulcer or growth. All the above findings suspicious for oral precancer on screening evaluation will be referred for further diagnostic evaluation by medical officers.

Control Arm:

No Active Intervention will be given in the control arm, but will distributed tobacco awareness pamphlets in local languages. Only base line and end line survey assessment will be done.

Training as tobacco cessation counselors & Development of Module.

1. Recruitment and training of staff This involves the recruitment of project personnel and their training. Training would involve the theoretical and practical teaching of questionnaire/survey as well modular training for tobacco cessation counseling to the project personnel.
2. Preparation of resource materials and questionnaire formats Resource materials would include training module for tobacco use prevention and tobacco cessation techniques with Individual and Group therapy sessions with pamphlets outlining the harmful effects of tobacco.

Outcome measures

The two outcome measures used from the survey questionnaire were 'ever use' and 'current use' of tobacco at baseline and endline. 'Ever users' were those who had consumed tobacco in any form in their life time. 'Current users' were those who had consumed tobacco in any form in the past one week. Current use at baseline and endline were compared to calculate the 'quit rate' and 'rate of fresh uptake'. Quit rate of tobacco use among the communities will be estimated as the proportion of workers who become non-users at endline from among those who were current users in the baseline survey. Rate of fresh uptake will be estimated as the proportion of workers who reported themselves as ever users or current users at endline from among those who were never users at the baseline survey.

Data Management and Analysis

Data will be entered and analyzed using SPSS version 18.3 The trial data will be analyzed on an intention to treat basis and the participants will be included in the final analysis irrespective of whether or not they could be followed up in all subsequent visits. Self reported history will be taken as the main criteria to assess outcome of tobacco cessation. Multivariate analysis will be performed to identify the factors promoting the use of tobacco and quitting tobacco. The tobacco quit rates will be calculated as percentages. The post intervention changes in the KAP of employees will be compared to the pre-intervention KAP. Groups will be compared using non-parametric statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate
2. All workers employed in each of the listed zari units.
3. Who are willing to give informed consent.

Exclusion Criteria:

1. Who are NOT willing to give informed consent.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Tobacco Quit Rate | 12 Months
  Tobacco quit rates in moderate intensity behavioural intervention, low intensity behavioral intervention and control group will be compared at the end of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila A Pimple, Professor, Principal Investigator — Tata Memorial Hospital; Gauravi A Mishra, Assoc Prof, Principal Investigator — Tata Memorial Hospital; Parishi Majmudar, MSW, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- See also: Tata Memorial Centre, Mumbai Official website — https://tmc.gov.in